CLINICAL TRIAL: NCT04840030
Title: Effectiveness of a Lifestyle Multidomain Intervention to Prevent Cognitive Decline in the Basque Country. GOIZ ZAINDU Gipuzkoa - CITA GO-ON Study
Brief Title: Preventing Cognitive Decline: The CITA GO-ON Multi-domain Intervention Study
Acronym: CITA GO-ON
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion CITA-alzheimer (Other)
Collaborators: Biogipuzkoa Health Research Institute (Other); University of the Basque Country (UPV/EHU) (Other); Achucarro Basque Center For Neuroscience (Unknown); NavarraBiomed Biomedical Research Center (Other); Basque Culinary Center Fundazioa (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Mikel Tainta, Principal Investigator, Fundacion CITA-alzheimer
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Go-on_studyprotocol_v3_apr20
Record Dates: First submitted 2021-03-26; First posted 2021-04-09 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Dementia; Cognitive Decline; Prevention; Life Style; Risk Factor, Cardiovascular; Diet Habit; Cognitive Intervention; Behavioral Intervention
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: The Gipuzkoa GOIZ ZAINDU - GO-ON study is a two year randomized, controlled trial to evaluate the effectiveness of multi-component lifestyle and dementia risk factor intervention in preventing cognitive decline in older adults with cognitive frailty.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard health advice (SHA-control) (No Intervention): The participant will receive verbal information of risk factors and information, reassessment, and written materials regarding approved recommendations on active and healthy aging on topics such as diet, physical activity, cognitive training as well as risk factor control following the state of the art and published guidelines by the Department of Health of the Basque Government/ Basque Country Public Health System (Osakidetza) and the WHO (Guidelines for risk reduction of cognitive decline and Dementia and the "Guidance on person-centered assessment and pathways in primary care - ICOPE"). Participants in this group will receive the best standard health care from their primary care and specialist health teams according to already established routines as well as usual social services assessments and care as needed.
- Multidomain intervention (MM-Int) (Experimental): Participants in this group will receive the same verbal and written recommendations as to the ones in the SHA-Control group but then they will perform a 2 year structured program with periodic individual and group visits regarding 1) Risk factor control (vascular factors, polypharmacy); 2) Cognitive training, 3) Physical activity, 4) Dietary changing program and 5) emotional counseling and social engagement.
  Interventions: Behavioral: Multimodal intervention (MM-int)

INTERVENTIONS:
Behavioral: Multimodal intervention (MM-int) — 1. Cognitive intervention objective: To enhance cognitive functioning and incorporate daily habits and routines that are cognitively stimulating
  2. Socio-emotional intervention objective: • Promote socio-emotional skills associated with awareness, communication and regulation of emotions in late life.
  3. Nutritional intervention objective: To improve eating habits of participants to be based on the Mediterranean Dietary pattern by an educational program
  4. Physical activity intervention objective: To improve aerobic capacity y, decrease the risk of falls, and improve static and dynamic balance.
  5. Risk factors and comorbidities monitoring intervention: quarterly scheduled visits for a cardiovascular risk factors check-up and review active medication
  Arms: Multidomain intervention (MM-Int)

SUMMARY:
The GOIZ ZAINDU Gipuzkoa - GO - ON Study is an intervention trial to evaluate the efficacy of dementia prevention strategies in cognitively frail people. It is a large-scale randomized controlled trial in over 1000 older adults between 60 and 85 years old with increased CAIDE risk score (≥6), non-demented but with low performance in at least one of three brief cognitive tests. Participants will be randomized to receive standard health advice (SHA-control) or a multidomain intervention (MM-Int) consisting of 1) Risk factor control (vascular factors, polypharmacy); 2) Cognitive training, 3) Physical activity, 4) Dietary changing program, and 5) emotional counseling and social engagement.

The primary aim is to demonstrate a 20% reduction in the proportion of subjects who decline in their NTB performance (z score) after 24 months in the intervention group compared to the controls.

Secondary aims include: 1) Analyze cost-effectiveness; 2) Show a beneficial effect of the intervention on functional abilities, quality of life, and depressive and anxiety symptoms; 3) Investigate the impact of a lifestyle intervention on aging. In this sense, biological samples and neuroimaging studies will be collected to allow exploratory investigations on aging mechanisms, amyloid imbalance, tau pathology, epigenetics, neuroinflammation, vascular dysfunction, lipid dysregulation, white matter disintegration, cognitive and brain reserve.

This protocol is participant-centered, empowering citizens since the recruitment process to gain access to knowledge about their dementia risk status via web or by phone and then decide to participate. Intervention activities have also taken into account participants' perspective with the design of easy-to-use and appealing activities (e.g., using a self-administered at-home physical activity program such as VIVIFRAIL© and EXERCITA© cognitive training materials that have been developed, taking into account the Basque Country population's cultural, linguistic and educational particularities; and diet and nutritional workshops with famous chefs to learn innovative and attractive healthy recipes).

The GO-ON trial may shed light on the tools that people need to fulfill the expectation of an active, healthy dementia-free aging. These include digital tools that in the COVID19 pandemic have shown to be effective in removing distance barriers. GO-ON uses them to give support and expand the possibilities to clinical assessment settings and intervention delivery. The digital part of the intervention may expand preventive actions to small rural areas, including digital socialization.

GO-ON Study, which starts in summer 2021, is the first large-scale lifestyle intervention trial in Southern Europe that takes part in the WORLDWIDE FINGERs network and will help answer whether the FINGER results can be replicated. The intervention design has been made on the basis that if proven to be efficacious, it may be easily applied at a Public System-level to guarantee a rapid and easy translation of research results to Primary Care settings and people homes.

ELIGIBILITY:
Inclusion Criteria:

1. People between 60-85 years old, willing to participate and comply with all the study evaluation and intervention procedures.
2. With a CAIDE dementia Risk score ≥ 6
3. Below-than-expected cognitive performance in at least one of three brief cognitive tests:

   * Fototest score ≤ 35
   * Memory Alteration Test -T@M score ≤40
   * Cognitive complaints as compared with a previous subjective performance - defined by a Cognitive Change Index - self-report version score >=20 on the first 12 (episodic memory) items to assist with defining Subjective Cognitive Decline (SCD) (Risacher et al. 2017).

Exclusion Criteria:

Exclusion criteria are conditions that may affect the achievement of study objectives and procedures or clinical diagnoses that by themselves compromise participant's cognitive performance or compliance with study procedures. They include:

1. Inability to perform a neuropsychological evaluation or a cognitive stimulation program (sensory limitation, mental retardation, illiteracy)
2. Barthel index < 90.
3. Geriatric Depression Scale ≥ 9
4. Dementia or Moderate Cognitive impairment (MMSE < 20).
5. Presence of any neurological, psychiatric or systemic disease that produce cognitive impairment or dementia including, but not limited to, Huntington's disease, multiple sclerosis, Parkinson's disease, Down syndrome, alcohol abuse or active drugs, or major psychiatric disorders including ongoing major depression, schizophrenia or bipolar or schizoaffective disorder.
6. Unstable ischemic cardiopathy, uncontrolled heart arrhythmia, thromboembolic disease in the last year. Moderate cardiorespiratory insufficiency (including Class III or IV congestive heart failure, clinically significant aortic stenosis, cardiac arrest history, or uncontrolled angina). Currently receiving physical therapy or cardiopulmonary rehabilitation.
7. Large vessel stroke in the past two years
8. History of transient ischemia attack (TIA) or small vessel stroke in the last 6 months
9. Any cerebrovascular accident with significant residual effects on cognition or functional autonomy.
10. History within the last 2 years of treatment for primary or recurrent malignant disease, excluding non-melanoma skin cancers, resected cutaneous squamous cell carcinoma in situ, basal cell carcinoma, cervical carcinoma in situ, or situ prostate cancer with normal prostate-specific antigen posttreatment
11. Recent (< 3 months) bone fracture.
12. History of hip fracture, joint replacement, or spinal surgery in the last 6 months
13. Clinically significant abnormalities in laboratory blood tests as per judgment of the site Study Clinician
14. Any conditions affecting safe engagement in the intervention in the judge of the study investigators.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1094 (Estimated)
Dates: Start 2021-12-03 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Global Cognitive performance | up to 2 years
  Cognitive performance will be assessed with the Neuropsychological Test Battery modified (NTBm) (Harrison J. et aet al.ch Neurol 2007).
  The NTBm consists of 9 validated components:NTBm Cognitive global, executive function, memory, processing speed scores will be obtained. Composite cognitive z-scores based on the results from all single tests will be calculated. Single z-scores will be calculated using baseline mean and standard deviations of the study sample and, for each composite score, single z-scores will be averaged. Higher scores suggest better performance.

SECONDARY OUTCOMES:
Performance in each cognitive domain | up to 2 years
  NTBm Cognitive global, executive function, memory, processing speed scores will be obtained. Composite cognitive z-scores based on the results from all single tests will be calculated. Single z-scores will be calculated using baseline mean and standard deviations of the study sample and, for each composite score, single z-scores will be averaged. Higher scores suggest better performance.
  b. Change in specific cognitive domains will be assessed by the difference in pre-and postintervention scores in episodic memory, executive function and processing speed and visuospatial function z-scores.
Incremental Cost-Utility Ratio (ICUR) | up to 2 years
  To estimate the cost-effectiveness of the intervention program the Incremental Cost-Utility Ratio (ICUR) between muntidomain intervention group and regular health advice group.
  The incremental cost-utility ratio (ICUR) will be estimated by dividing incremental cost (Ca-Cb) by incremental utility (Ua-Ub). The time horizon was the patient's lifetime. A 3% discount rate will be applied to costs and effectiveness. Since the main economic impact of dementia is related to the care required as patients become dependent, a societal perspective will be used.
Amsterdam questionnaire for Instrumental Activities of Daily Living (A-IADL-Q) | up to 2 years
  The Amsterdam IADL Questionnaire (A-IADL-Q) is an adaptive and computerized questionnaire designed to assess impairments in instrumental activities of daily living (IADL) in (early) dementia. The questionnaire is completed by a caregiver, such as a relative or friend. (Sikkes SA et al. 2012).
Change in perceived Quality of life - EQ-D-5L scale | up to 2 years
  The EQ-5D-5L (Herdman M. et al. 2011) essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Depressive and anxiety sympthoms. Hospital Anxiety and Depression Scale (HADS) | up to 2 years
  HADS was originally developed by Zigmond and Snaith (1983) and is commonly used to determine the levels of anxiety and depression that a person is experiencing. The HADS is a fourteen-item scale that generates: Seven of the items relate to anxiety and seven relate to depression.
Change in cognitive performance in different groups of patients with the same APOE status | up to 2 years
  To assess whether differences between intervention groups concerning the primary and secondary cognitive outcomes vary among subgroups defined by APOE status as a genetic condition.

CONTACTS AND LOCATIONS:
Overall Officials: Mikel Tainta, MD, Principal Investigator — Principal Investigator; Pablo Martinez-Lage, MD PhD, Study Chair — Scientific Director
Locations (1):
- CITA-alzheimer, Donostia / San Sebastian, Gipuzkoa, Spain

IPD SHARING:
Plan to Share IPD: Yes
Access to research raw data will be available after request. Following the foundational principles of data harmonization from the Worldwide FINGERs network, data might be shared after assuring participants' confidentiality and privacy, with WWFINGERs leaders from Karolinska Institute.

REFERENCES:
- [Background] Ngandu T, Lehtisalo J, Solomon A, Levalahti E, Ahtiluoto S, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H, Kivipelto M. A 2 year multidomain intervention of diet, exercise, cognitive training, and vascular risk monitoring versus control to prevent cognitive decline in at-risk elderly people (FINGER): a randomised controlled trial. Lancet. 2015 Jun 6;385(9984):2255-63. doi: 10.1016/S0140-6736(15)60461-5. Epub 2015 Mar 12. PMID 25771249